CLINICAL TRIAL: NCT01295489
Title: A Study of the Local and Systemic Effects of Intraperitoneal Chemotherapy in the Treatment of Previously-Untreated, Invasive Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma
Brief Title: Biomarkers in Patients With Previously Untreated Invasive Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0271; NCI-2011-02871 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000695260; GOG-0271 (Other: NRG Oncology); GOG-0271 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Fallopian Tube Carcinoma; Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

GROUPS / COHORTS (2):
- Group A (IP catheter removed): Archival formalin-fixed, paraffin-embedded tumor (collected during previous surgery), peritoneal fluid, peritoneal wash, and blood (for cell, plasma, and serum isolation) samples are collected before course one and blood (for cell, plasma, and serum isolations) is collected before courses two and three for translational research.
  Interventions: Other: Laboratory Biomarker Analysis
- Group B (IP catheter in place): Archival formalin-fixed, paraffin-embedded tumor (collected during previous surgery), peritoneal fluid, peritoneal wash, and blood (for cell, plasma, and serum isolation) samples are collected before course one and peritoneal fluid, peritoneal wash, and blood (for cell, plasma, and serum isolations) before courses two and three for translational research.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies biomarkers in patients with previously untreated invasive ovarian epithelial, fallopian tube, or primary peritoneal cancer. Studying samples of tumor tissue, peritoneal cavity fluid, and blood from patients receiving chemotherapy directly into the abdominal cavity (intraperitoneal) may help doctors learn more about the effects of intraperitoneal chemotherapy on cells. It may also help doctors identify and learn more about biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of obtaining peritoneal fluid, peritoneal washings, and peripheral blood in patients receiving intraperitoneal (IP) chemotherapy for ovarian cancer at multiple institutions.

II. Assess the recovery and viability of peripheral blood mononuclear cells and immune cell subsets in peritoneal fluid and washings.

III. Assess the amount of peritoneal fluid that can be obtained pre-treatment and at specified time points during the course of IP chemotherapy.

IV. Quantify the type and number of cells in peritoneal fluid, peritoneal washings, and blood recovered from women before and during treatment with platinum and taxane based IP chemotherapy.

V. Determine the levels of immunomodulatory cytokines in peritoneal fluid, peritoneal washings, and blood recovered from women before and during treatment with platinum and taxane based IP chemotherapy.

VI. Generate exploratory information on the impact of platinum and taxane based IP chemotherapy on immunomodulatory cytokines and tumor-associated alterations in cell phenotypes of peritoneal fluid, peritoneal washings, and blood.

VII. To determine the feasibility of obtaining peritoneal fluid, peritoneal washings, and peripheral blood in patients receiving intravenous (IV) chemotherapy for ovarian cancer at multiple institutions (limited to patients that receive an IP catheter at the time of surgery and the catheter is left in by the investigator, but are subsequently treated with IV chemotherapy).

VIII. Assess the amount of peritoneal fluid that can be obtained pre-treatment and at specified time points during the course of IV chemotherapy.

IX. Assess the recovery and viability of peripheral blood mononuclear cells and immune cell subsets in peritoneal fluid and washings.

X. Quantify the type and number of immune cells in peritoneal fluid, peritoneal washings, and blood recovered from women before and during treatment with platinum and taxane based IV chemotherapy.

XI. Determine levels of immunomodulatory cytokines in peritoneal fluid, peritoneal washings, and blood recovered from women before and during treatment with platinum and taxane-based IV chemotherapy.

XII. Generate exploratory information on the impact of platinum and taxane based IV chemotherapy on immunomodulatory cytokines tumor-associated alterations in cell phenotypes of peritoneal fluid, peritoneal washings, and blood.

XIII. Explore whether there is a relationship between immune cell populations measured in peripheral blood, peritoneal fluid, and peritoneal washings AND immune cell subsets measured by immunohistochemistry in archival formalin-fixed, paraffin-embedded tumor tissue.

OUTLINE: Patients are assigned to a group based on which arm of treatment they are randomized to receive on Gynecologic Oncology Group (GOG)-0252.

GROUP A (IP CATHETER REMOVED): Archival formalin-fixed, paraffin-embedded tumor (collected during previous surgery), peritoneal fluid, peritoneal wash, and blood (for cell, plasma, and serum isolation) samples are collected before course one and blood (for cell, plasma, and serum isolations) is collected before courses two and three for translational research.

GROUP B (IP CATHETER IN PLACE): Archival formalin-fixed, paraffin-embedded tumor (collected during previous surgery), peritoneal fluid, peritoneal wash, and blood (for cell, plasma, and serum isolation) samples are collected before course one and peritoneal fluid, peritoneal wash, and blood (for cell, plasma, and serum isolations) before courses two and three for translational research.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on GOG-0252
* Patients must have an IP catheter placed prior to initiating platinum and taxane-based chemotherapy on GOG-0252
* Patients must have signed an approved informed consent for specimen collection and participation in this translational research study

Exclusion Criteria:

* Patients who are not enrolled on GOG-0252
* Patients who have not had an IP catheter placed prior to initiating platinum and taxane-based IP chemotherapy on GOG-0252
* Patients who did not sign an approved informed consent for specimen collection and participation in this translational research study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2011-03; Primary Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Amount of peritoneal fluid obtained during each attempted extraction of peritoneal fluid or washing | Up to 1 year
Presence of immune cells measured by immunohistochemistry in archival formalin-fixed, paraffin-embedded tumor tissue | Up to 1 year
  The staining intensities of immune cells detected in immunohistochemically stained paraffin tissue will be described using descriptive statistics such as the median, 1st and 3rd quartiles of staining intensities. Spearman's correlation coefficient will be used to assess associations between these intensities and the cell counts obtained from pre-treatment peripheral blood and peritoneal fluids. Boxplots or scattergrams will be used to display these data.
Quantity of each type of immune cells identified in the peritoneal fluid or washings specimens | Up to 1 year
  A Wilcoxon signed rank test will be used to evaluate the null hypothesis that the expectation of the pretreatment cell counts is equal to the expectation of the post-treatment cell count. Descriptive statistics such as the mean, variance, median, 1st and 3rd quartiles as well as the spearman correlation between pre- and post- treatment cell counts will be reported for each cell type. Boxplots or scattergrams will be used to display the results. The mean, variance and quartiles of the amount of fluid recovered from pre-treatment and post-treatment samples will also be reported.
Quantity of each type of mononuclear cells in peripheral blood | Up to 1 year
  The number and type of mononuclear cells in peripheral blood will be described using descriptive statistics such as the median, 1st and 3rd quartiles. Spearman's correlation coefficient will be used to assess associations between pre- and post- treatment values. Boxplots or scattergrams will be used to display these data. A Wilcoxon signed rank test, that involves the patients' pre- and post- treatment measurements, will be used to evaluate the null hypothesis that these cell counts are unchanged by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, Principal Investigator — NRG Oncology
Locations (9):
- United States (9):
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Billings Clinic Cancer Center, Billings, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island